CLINICAL TRIAL: NCT03369873
Title: Effectiveness of Nursing Orientation for the Reduction of Anxiety and Stress of Patients That Waiting Cardiac Catheterization: Randomized Clinical Trial.
Brief Title: Effectiveness of Nursing Orientation for the Reduction of Anxiety and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Juliana de Lima Lopes, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UNIFESP30
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Coronary Syndrome
Keywords: cardiac catheterization; anxiety; stress; nursing orientation
MeSH Terms: conditions — Angina, Unstable; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The patients were randomized to one of two groups (control or intervention), according to the sequence determined by the Random System
Who Masked: Outcomes Assessor
Masking Description: The profissional that evaluated the patients, was not informed if the patients were of the control or intervention group. The outcomes assessor was not informed if the group 1 and 2 was control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing Orientation with guidance manual (Experimental): The patients received the nursing orientation with validated guidance manual of cardiac catheterization.
  Interventions: Other: Guidance Manual
- Routine Nursing Orientation (No Intervention): The patients received the routine nursing orientation about cardiac catheterization.

INTERVENTIONS:
Other: Guidance Manual — The intervention group received of nursing orientation using a validated guidance manual about cardiac catheterization.
  Other Names: Routine Orientation
  Arms: Nursing Orientation with guidance manual

SUMMARY:
This study´s objective was to identify the effectiveness of nursing orientation for the reduction of anxiety and stress of patients that was waiting cardiac catheterization. Method. This is a randomized clinical trial. The sample consisted of patients that was waiting cardiac catheterization who were divided into two groups: intervention group (patients who received nursing orientation with a validated guidance manual about this procedure) and control group (patients who received the routine nursing orientation). The primary end points were the anxiety and stress, which was evaluated in two moments (before and after the nursing orientation). The State Anxiety Inventory (STAI-state) was used to assess anxiety and the Perceived Stress Scale (PSS-10) was used to assess stress. Prior to the collection, the research project was submitted to the Research Ethics Committee and the data was collected after its approval.

DETAILED DESCRIPTION:
This study´s objective was to identify the effectiveness of nursing orientation for the reduction of anxiety and stress of patients that was waiting cardiac catheterization. Method. This is a randomized clinical trial. The sample consisted of patients that was waiting cardiac catheterization who were divided into two groups: intervention group (patients who received nursing orientation with a validated guidance manual about this procedure) and control group (patients who received the routine nursing orientation). The subjects were consulted about the desire to participate, and those who agreed, signed the consent form. The patients were randomized to one of two groups (control or intervention), according to the sequence determined by the Random System. Randomization was carried out by a teacher who did not participate of any phase of this study. After randomization, the patients were instructed how to fill out the instruments. The primary end points were the anxiety and stress, which was evaluated in two moments (before and after the nursing orientation). The State Anxiety Inventory (STAI-state) was used to assess anxiety and the Perceived Stress Scale (PSS-10) was used to assess stress. Subsequent to this first evaluation, the patients, both in the control group and in the intervention group, received the intervention by another profissional. After the patients were evaluated about anxiety and stress. Prior to the collection, the research project was submitted to the Research Ethics Committee and the data was collected after its approval.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years
* Literate
* Stable patients in Killip I and II
* Maximum 79 years

Exclusion Criteria:

* Hemodynamic instability
* Precordial pain
* Patients who undergo emergency cardiac catheterization
* Patients with visual deficit and / or with some alteration of the level of consciousness
* Patients using benzodiazepine, anxiolytic and / or herbal medicines
* Situations that patient received orientation about the procedure prior to initiation of the current hospitalization survey and / or when reporting that they do not wish to receive information.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change from score of anxiety and stress | The patients were followed for one day
  The anxiety and stress were evaluated using the State Anxiety Inventory (STAI-state) and the Perceived Stress Scale (PSS-10), immediately before and after interventions. The STAI -state consists of 20 items, with Likert responses ranging from 1 (Absolutely not) to 4 (Very High), obtaining values from 20 to 80 points, that the higher the score, the greater the patient's anxiety. Anxiety was categorized as follows: low anxiety (20-34 points), moderate anxiety (35-49 points), high anxiety (50-64 points) and very high anxiety (65-80 points). The PSS-10 has 10 items, whose score varies from 0 to 40 points, and the higher the scores, the greater the perceived stress of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana de L Lopes, PhD, Study Director — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: No
We not plan to make individual participant data avaiable to other researchers.

REFERENCES:
- [Background] Peterson JC, Link AR, Jobe JB, Winston GJ, Marina Klimasiewfski E, Allegrante JP. Developing self-management education in coronary artery disease. Heart Lung. 2014 Mar-Apr;43(2):133-9. doi: 10.1016/j.hrtlng.2013.11.006. Epub 2013 Nov 25. PMID 24373484
- [Background] Reis RS, Hino AA, Anez CR. Perceived stress scale: reliability and validity study in Brazil. J Health Psychol. 2010 Jan;15(1):107-14. doi: 10.1177/1359105309346343. PMID 20064889
- [Background] Wu KL, Chen SR, Ko WC, Kuo SY, Chen PL, Su HF, Chang WY. The effectiveness of an accessibility-enhanced multimedia informational educational programme in reducing anxiety and increasing satisfaction of patients undergoing cardiac catheterisation. J Clin Nurs. 2014 Jul;23(13-14):2063-73. doi: 10.1111/jocn.12469. Epub 2013 Dec 27. PMID 24372795
- [Derived] Murakami L, Rua ES, Santos VB, Lopes JL. Effectiveness of educational intervention with manual for anxiety and stress reduction: controlled clinical trial. Rev Bras Enferm. 2022 Sep 5;75Suppl 3(Suppl 3):e20210757. doi: 10.1590/0034-7167-2021-0757. eCollection 2022. English, Portuguese. PMID 36074457